CLINICAL TRIAL: NCT00332215
Title: Inhaled Sodium Pyruvate for the Treatment of Cystic Fibrosis. A Phase I, Double Blind, Placebo Controlled, Safety Study.
Brief Title: A Phase I Study of Inhaled Sodium Pyruvate for the Treatment of Cystic Fibrosis.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Dr. Milla has left University of Minnesota. The study is no longer being conducted at this site.
Sponsor: University of Minnesota (Other)
Collaborators: Cellular Sciences, inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0511M77511; CSI-N115-I-010-01
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Antioxidants; Inhalational therapy; Induced sputum; Airway inflammation
MeSH Terms: conditions — Cystic Fibrosis

INTERVENTIONS:
Drug: Inhaled Sodium Pyruvate

SUMMARY:
The primary objective of this study is to assess the safety of inhaled sodium pyruvate in people with Cystic Fibrosis (CF). Further, to determine whether inhaled sodium pyruvate will improve lung function, as determined by FEV1, or reduce inflammatory markers in induced sputum of people with CF.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a disease that causes airway blockage and infection that damages the lung. The lungs of CF patients are frequently loaded with inflammatory cells, damaging proteins and oxidants. Oxidants are molecules that contain oxygen and are capable of disrupting cells and tissue. The CF protein is involved in the transport of the important antioxidant glutathione (GSH). Antioxidants are molecules that block oxidants and render them inactive. The absence of this protection in the airways makes them prone to damage from oxidants. Sodium pyruvate is part of the body's natural anti-oxidant defense system. Sodium pyruvate reacts directly with oxygen radicals to neutralize them and increases cellular levels of glutathione.

The purpose of this study is to investigate the safety and tolerability of 3 different single dose levels of sodium pyruvate administered via a nebulizer to persons with CF lung disease.

This will be a phase I study with 3 stages. In the first stage subjects will receive one of 3 possible doses of the active drug only once. In the second stage subjects will receive 2 doses of the active drug 12 hours apart. In the third stage subjects will receive either active drug or placebo every 12 hours for 4 weeks.

For stage 1 subjects will come to the University of Minnesota's General Clinical Research Center (GCRC) for a screening visit. They will return to the GCRC 1 to 7 days later for a baseline assessment that will be followed by study drug administration. The subject will be observed for 4 hours and safety parameters will be obtained.

For stage 2 subjects will come to the GCRC for a screening visit. They will return to the GCRC 1 to 7 days later for a baseline assessment that will be followed by study drug administration. Safety parameters will be obtained for the following 4 hours. 12 hours after the first dose was given the subject will receive a second dose and safety parameters will again be obtained over the next 4 hours.

For stage 3 subjects will come to the GCRC for a screening visit. They will return to the GCRC 1 to 7 days later for a baseline assessment that will be followed by study drug administration. Safety parameters will be obtained for the following 4 hours. The subject will be sent home to continue on study drug every 12 hours for the following 4 weeks. The subject will be asked to return to the GCRC once a week for safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CF using Cystic Fibrosis Foundation criteria.
* FEV1 >40% predicted
* Colonization with Pseudomonas aeruginosa - (>= 2 positive cultures over past 12 months)
* >18 years of age
* Stable respiratory status without dyspnea at rest
* Non-smoker
* Able to perform sputum induction

Exclusion Criteria:

* Severe CF lung disease with an FEV1 of <40% predicted
* Lung disease not CF related
* Positive culture for Burkholderia cepacia over previous 2 years
* Active allergic bronchopulmonary aspergillosis
* Clinically significant cardiac disease
* Pregnancy
* Females of child bearing age not using contraception
* Females lactating
* <18 years of age
* Systemic steroid treatment within 1 month
* Hospitalization within 3 months due to airway disease
* Immunotherapy
* Changes in respiratory medication use within 1 month
* New medications within 1 month
* Administration of any investigational drug or device within 28 days of visit 1 or within 6 half-lives of the investigational drug (whichever is longer).
* History of significant (>60 cc) hemoptysis within 1 year
* Poorly controlled insulin dependent diabetes mellitus
* Acute respiratory illness within 1 month
* Use of tobacco products or recreational drugs
* History of adverse reaction to sputum induction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2006-02

PRIMARY OUTCOMES:
The primary outcome variable is the assessment of safety of inhaled sodium pyruvate in subjects with CF.Subjects will be evaluated for the presence of symptoms and safety laboratory measurements.

SECONDARY OUTCOMES:
The secondary outcome variable is the determination of improvement in lungs of CF subjects as determined by measurement of FEV1 and measurement of inflammatory markers in induced sputum.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E Milla, MD, Principal Investigator — University of Minnesota; Joanne L Billings, MD, MPH, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota General Clinical Research Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] O'Donnell-Tormey J, Nathan CF, Lanks K, DeBoer CJ, de la Harpe J. Secretion of pyruvate. An antioxidant defense of mammalian cells. J Exp Med. 1987 Feb 1;165(2):500-14. doi: 10.1084/jem.165.2.500. PMID 3102672
- [Background] Votto J, Bowen J, Metersky M, Thrall R. Effect of Inhaled Sodium Pyruvate in Patients with Mild Bronchial Asthma. Am J Resp Crit Care Med 2001, 163 (5S):A860.